CLINICAL TRIAL: NCT05979402
Title: Effectiveness of Pressure Wound Prevention Training for the Relatives of Palliative Care Patients: A Randomized Controlled Trial
Brief Title: The Effect of Pressure Ulcer Education on the Knowledge Level of the Relatives of the Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Lutfiye Nur Uzun, PhD, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AIBU-HEM-UZUN-004
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Pressure Ulcer; Caregiver Education; Palliative Care
MeSH Terms: conditions — Pressure Ulcer | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled study with experimental and control groups consisting of pre-test and post-test
Who Masked: Outcomes Assessor
Masking Description: Outcome evaluations will be conducted by a researcher blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Face-to-face pressure ulcer training will be given to the relatives of the patients in the training group in the determined common time period. The presentation and pressure ulcer content prepared during the trainings will be conveyed by the researcher in two 30-minute sessions using lectures, example events and question-answer techniques.
  Interventions: Other: Training group Face-to-face pressure ulcer training
- Control group (Active Comparator): Participants in the control group will not be interfered with by the researcher during the research. They will receive routine in-clinic training given by nurses.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Training group Face-to-face pressure ulcer training — Face-to-face presure ulcer training
  Arms: Training group
Other: Control group — No intervention
  Arms: Control group

SUMMARY:
The purpose of this randomized controlled trial, which included pretest and posttest, was to examine the effectiveness of pressure ulcer prevention and care education given to caregivers of patients treated in a palliative care clinic.

The key questions it aims to answer are:

* Does the routine clinical training given in the palliative care clinic have an effect on the knowledge level of patients' relatives about pressure ulcers?
* Does the pressure ulcer education given to the relatives of patients treated in the palliative care clinic have an effect on the level of knowledge about pressure ulcers?

Participants will participate in an educational activity on pressure ulcers. Researchers will compare whether pressure ulcer training given to palliative care patient relatives is effective compared to routine service training with lecture, question-answer and presentation method.

DETAILED DESCRIPTION:
One-to-one interviews will be conducted with the relatives of the patients in the experimental and control groups, and the appropriate time frame for the clinical operation will be determined. Participants will be informed about the study at the time determined jointly with the companions and at the appropriate place for the clinic.

Personal Information Form and Pressure Ulcer Information Test will be distributed and collected as a pre-test to the participants in the control group. The participants in the control group will not receive any educational intervention by the researcher until the day of discharge. This group will receive routine clinical training given only in the hospital. Training of patients and their relatives in clinics continues with the principle of "Do-Watch-Check". This is how nurses conduct their routine clinical training. The Pressure Ulcer Information Test will be distributed and collected as a post-test to the control group on the day of the patients' discharge.

Personal Information Form and Pressure Ulcer Information Test will be distributed and collected as a pre-test to the participants in the experimental group. In addition to the training given to the participants in the experimental group with the routine "Do-Watch-Check" principle in the clinic, face-to-face pressure ulcer training will be given by the researchers on the day of discharge. The presentation about the pressure ulcer will be given by the researchers in two periods of 30 min + 30 minutes using lectures, case studies and question-answer techniques. Opinions were received from three field experts regarding the validity of the training content of the pressure ulcer topic (CGI: 1.00). The Pressure Ulcer Knowledge Test will be redistributed and collected as a final test on the day of discharge after completion of training.

ELIGIBILITY:
Inclusion Criteria:

* Those who agree to participate in the study
* Native Turkish,
* 18 years and over
* Able to read and write

Exclusion Criteria:

* Who refused to participate in the study
* Native language is not Turkish
* Illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Pressure ulcer information of palliative care patients' relatives: First test | Just before training
  "Pressure Ulcer Knowledge Test" is a test prepared by researchers in line with the literature and sent to three expert academicians to ensure content validity. Pressure Ulcer Knowledge Test is a 3-point Likert-type questionnaire consisting of 17 questions coded as true, false, I don't know. Five of the questions in the test were designed to be scored reversely and 12 of them were scored straight. The score to be taken from the test is between 0-17. A high score indicates that the relatives of the patients have a high level of knowledge about pressure ulcers, and a low score indicates a low level of knowledge.

SECONDARY OUTCOMES:
Pressure ulcer information of palliative care patients' relatives: Second test | Immediately after training
  "Pressure Ulcer Knowledge Test" is a test prepared by researchers in line with the literature and sent to three expert academicians to ensure content validity. Pressure Ulcer Knowledge Test is a 3-point Likert-type questionnaire consisting of 17 questions coded as true, false, I don't know. Five of the questions in the test were designed to be scored reversely and 12 of them were scored straight. The score to be taken from the test is between 0-17. A high score indicates that the relatives of the patients have a high level of knowledge about pressure ulcers, and a low score indicates a low level of knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfiye Nur Uzun, PhD, Principal Investigator — Bolu Abant İzzet Baysal University Faculty of Health Sciences Nursing Department; Hümeyra Hançer Tok, PhD, Principal Investigator — Bolu Abant İzzet Baysal University Faculty of Health Sciences Nursing Department

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.

REFERENCES:
- [Derived] Hancer Tok H, Uzun LN. Pressure ulcer prevention: family caregiver training effectiveness. BMJ Support Palliat Care. 2024 Dec 25;15(1):72-78. doi: 10.1136/spcare-2023-004711. PMID 38253489